CLINICAL TRIAL: NCT06314477
Title: Effect of CPAP Treatment on Asthma Control in Patients With Severe Uncontrolled Asthma and Obstructive Sleep Apnea: The ASTHMA-SLEEP Study
Brief Title: Effect of CPAP Treatment in Patients With Severe Uncontrolled Asthma: The ASTHMA-SLEEP Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Mireia Dalmases, Principal investigator, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HCB/2022/1204
Record Dates: First submitted 2024-02-25; First posted 2024-03-18 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Obstructive Sleep Apnea; Asthma
MeSH Terms: conditions — Sleep Apnea, Obstructive; Asthma | interventions — Continuous Positive Airway Pressure; Nutrition Assessment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conservative treatment (Active Comparator): Subjects allocated to this arm will receive hygienic and dietary measures counselling
  Interventions: Other: Hygienic and dietary advice
- CPAP treatment (Experimental): Subjects allocated to this arm will receive treatment with continuous positive airway pressure (CPAP)
  Interventions: Device: CPAP treatment

INTERVENTIONS:
Device: CPAP treatment — Subjects allocated to this arm will receive continuous positive airway pressure (CPAP)
  Arms: CPAP treatment
Other: Hygienic and dietary advice — Subjects allocated to this arm will receive hygienic and dietary counselling
  Arms: Conservative treatment

SUMMARY:
The aim of the study is to evaluate the impact of CPAP treatment on asthma control in patients with severe uncontrolled asthma and obstructive sleep apnea (OSA)

DETAILED DESCRIPTION:
Background: The prevalence of obstructive sleep apnea (OSA) is high in patients with severe uncontrolled asthma and can worsen asthma control. Previous observational studies demonstrated that CPAP treatment could improve control in patients with mild-moderate asthma. Nevertheless, there are no studies in patients with severe uncontrolled asthma.

Primary objective: To evaluate the impact of CPAP treatment on asthma control in patients with severe uncontrolled asthma and AOS.

Methodology: Multicenter, prospective, randomized, controlled clinical trial with parallel groups in subjects with severe uncontrolled asthma who are older than 18 years and without sleepiness (Epworth sleepiness scale score ≤10). All included subjects will undergo conventional polysomnography and those with an apnea-hypopnea index (AHI) ≥15/hour will be randomized in a 1:1 ratio to receive conservative treatment or conservative treatment plus CPAP. Monitoring will be carried out during12 months. Patients will be evaluated at inclusion, at 1 month, 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Diagnosis of severe uncontrolled asthma according to the criteria of the Spanish Asthma Management Guide (GEMA) or the Global Initiative for Asthma (GINA) and no hospitalizations the month prior to inclusion in the study.
* Apnea hypopnea rate greater than or equal to 15/hour
* Punctuation in the Epworth Sleepiness Scale ≤10
* Obtaining informed consent.

Exclusion Criteria:

* Previous treatment with CPAP
* Patient with central sleep apnea or Cheyne-Stokes respiration
* Other sleep disorders: narcolepsy, restless leg syndrome, chronic insomnia,
* Resistant hypertension
* Active Smoking
* Unstable comorbidities or medications may interfere with asthma control
* Pregnancy
* Any process that reduces life expectancy to <1 year,
* Any medical or social factor that may limit CPAP compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2023-12-27 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Asthma control questionnaire | 12 months
  To evaluate the impact of CPAP treatment on asthma control based on the Asthma control questionnaire (ACQ)
Asthma control test | 12 months
  To evaluate the impact of CPAP treatment on asthma control based on the Asthma control test (ACT)

SECONDARY OUTCOMES:
Lung function- forced expiratory volume in the first second (FEV1) in spirometry | 12 months
  To evaluate the impact of CPAP treatment on FEV1 (ml) on spirometry
Lung function-forced vital capacity (FVC) in spriometry | 12 months
  To evaluate the impact of CPAP treatment on FVC (ml) on spirometry
Prevalence of OSA in severe uncontrolled asthma | Baseline
  Determine the prevalence of OSA in patients with severe uncontrolled asthma
Inflammatory profile | Baseline and 12 months
  Plasma proteins from peripheral blood samples will be used to analyze an inflammatory panel using a high-throughput, multiplex immunoassay technology based on Proximity Extension Assays (PEA) at baseline and after CPAP treatment
Quality of life (Abbreviated Asthma Quality of life Questionnaire- mini-AQLQ questionnaire) | 12 months
  Study whether OSA ans its treatment affects quality of life in subjects with severe uncontrolled asthma based on the punctuation obtained in the mini-AQLQ questionnaire. Higher scores indicate better quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Mireia Dalmases, MD, Principal Investigator — Hospital Clinic
Locations (1):
- Hospital Clinic Barcelona, Barcelona, Spain, Spain

IPD SHARING:
Plan to Share IPD: Undecided